CLINICAL TRIAL: NCT01465126
Title: Collagen Type 4-related Nephropathies: From Alport to Thin Membrane Nephropathy. A Series of Cases Treated With Angiotensin Converting Enzyme Inhibitor
Brief Title: Enalapril in Collagen Type 4 Nephropathy
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Maria Helena Vaisbich, Principal Investigator, University of Sao Paulo
Other Study IDs: Registry Identifier
Record Dates: First submitted 2011-10-27; First posted 2011-11-04 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-11

CONDITIONS: Collagen Type-4 Nephropathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: Collagen IV-related nephropathies can lead to End Stage Renal Disease. Experimental studies have shown renin angiotensin aldosterone system blockade can reduce proteinuria and preserve renal function. In humans there is no proven treatment. Methods: This is a retrospective study of patients with Collagen IV-related nephropathies and proteinuria treated with enalapril analyzing the evolution of proteinuria and renal function, as well as predictive variables of progression to end stage renal disease. Outcome was creatinine clearance < 60 ml/min/1.73m2.

DETAILED DESCRIPTION:
Introduction Collagen IV-related nephropathies, caused by mutations in the three genes encoding collagen type IV of the basal membrane, represent a spectrum of phenotypes from Alport syndrome (AS) to thin basement membrane nephropathy (TBMN) (1). Subtypes are X-linked AS (XLAS) which corresponds approximately 80% of AS, autosomal recessive AS (ARAS), counting for 15% of AS, and the autosomal dominant forms, represented by autosomal dominant AS (ADAS, 5% of AS) and TBMN, which is believed to be present in 1% of the population (1).

Besides renal manifestations, these diseases can present cochlear and ocular abnormalities (2). However, the hallmark of Collagen IV-related nephropathies is hematuria. Proteinuria is detected during life, being a marker of disease progression. All males with XLAS develop proteinuria and, eventually, progressive renal insufficiency, which leads to end-stage renal disease (ESRD). Overall, an estimated 60% reach ESRD by age 30 years, and 90% by age 40 years (2). Approximately 12% of females with XLAS develop ESRD before age 40 years, increasing to 30% by age 60 years (3). Most individuals with ARAS develop significant proteinuria in late childhood or adolescence and ESRD before age 30 years. Progression to ESRD is slower in individuals with ADAS. Similarly, TBMN is characterized clinically by persistent microhematuria often observed in childhood. TBMN is rarely associated with extrarenal abnormalities and proteinuria. Hypertension and progression to ESRD are unusual (4).

Despite the severity of disease, the high rate of ESRD, and the increasing knowledge about genetics and diagnosis, there is currently no proven treatment to AS. So far, the therapeutic approach is limited to angiotensin-II (AII) blockade, blood pressure control and diet counseling. Angiotensin-converting enzyme inhibitors (ACEi) or angiotensin receptor blockers (ARB) are usually started once proteinuria appears but there is no clear evidence that such treatment alters the natural history of the disease in humans.

Our goal was to describe the evolution of a series of cases with Collagen IV-related nephropathies and proteinuria treated with enalapril, as well as predictive variables of progression to ESRD.

Patients and Methods This is a retrospective study of collagen IV-related nephropathies patients followed at Instituto da Criança - HCFMUSP from 1999 to 2010. All patients presented glomerular hematuria (erythrocyte dysmorphism and/or red blood cell cast in the urinary sediment) and proteinuria. In 16 of 19 cases the diagnosis was based on familial history and renal histology findings which showed negative immunofluorescence and the ultrastructural abnormalities of the glomerular basement membrane (GBM) showing TBMN (uniform or diffuse attenuation of the GBM without the typical lamellation and thickening that is seen in AS) or AS (defects in terms of alternating attenuation, splitting, lamellation, and thickening along the GBM). However, it is very difficult to discriminate between the initial stage of AS and TBMN. Three patients were not submitted to renal biopsy since the familial history and the renal histology of relatives were characteristics of the disease. Only adherent patients were included, which was based on presence in attendance and exams.

The patients visited the outpatient clinic at least once every 3 months and had at least 2 years of follow up. The following parameters were evaluated at baseline: age, renal function (serum creatinine, urea, and creatinine clearance according to Schwartz Formula) (5), 24 hour proteinuria, blood pressure and light and electron microscopy of the renal fragment.

In all patients, enalapril was employed as a RAAS blocker, observing benefits and side effects as hypotension symptoms and/or signs. Our protocol intends to reach a dose of 0.3 mg/kg/day.

The following parameters were also collected during follow up: serum creatinine and urea, 24 hour proteinuria and creatinine clearance estimated by stature (Schwartz Formula).

In this study hyperfiltration is defined as ≥ 145 ml/minute/1.73m2BS, based on Piepsz et al and Prestidge et al data (6,7).

Statistical analysis Mann-Whitney and chi-square (or Fisher) tests were used in the univariate analysis. For the analysis of the effect of enalapril on proteinuria during the first 2 years of treatment we have used a non-parametric repeated measures analysis (Friedmann´s test). We have analyzed the main predictive variables of CKD progression, by considering a creatinine clearance below 60 ml/min/1.73m2 as an outcome.

ELIGIBILITY:
Inclusion Criteria:

* age under 18 years old
* non-adherent to the exams and evaluations

Exclusion Criteria:

* creatinine clearance < 60 ml/minute/1.73m2BS

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Collagen type 4 nephropathies and proteinuria followed in Pediatric Nephrology Unit of Instituto da Criança - HCFMUSP
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2011-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
proteinuria | two years
  evaluate the proteinuria during two years of treatment with enalapril

SECONDARY OUTCOMES:
evaluate the creatinine clearance during treatment with enalapril | two years